CLINICAL TRIAL: NCT03704181
Title: Effect of Colchicine on Inflammation and Myocardial Fibrosis Assessed by Magnetic Resonance Imaging in Patients With Chagas' Heart Disease
Brief Title: Colchicine for Patients With Chagas´ Disease( B1 Stage)
Acronym: COACH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4436/16/102
Record Dates: First submitted 2018-09-27; First posted 2018-10-12 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2018-09

CONDITIONS: Chagas Disease; Colchicine Resistance
Keywords: fibrosis; Inflammation
MeSH Terms: conditions — Chagas Disease; Fibrosis; Inflammation | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- colchicine (Experimental): colchicine 0,5 milligram tablet by mouth every 12 hours, for 1 year
  Interventions: Drug: Colchicine 0.5 MG twice day for one year
- placebo (Active Comparator): placebo tablet by mouth every 12 hours, for 1 year
  pill manufactured to mimic coclchicine 0,5 mg tablet
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Colchicine 0.5 MG twice day for one year — placebo twice day for one year
  Other Names: placebo oral tablet
  Arms: colchicine
Drug: Placebo Oral Tablet — placebo twice day for one year
  Arms: placebo

SUMMARY:
This study evaluate the addition of colchicine in the treatment of patients with Chagas´disease.

Forty patients will receive colchicine while twenty patients will receive placebo

DETAILED DESCRIPTION:
Chagas disease is considered one of the main cause of dilated cardiomyopathy in Latin America. The histopathological characteristics of Chagas' disease are the presence of myocarditis, destruction of heart fibers, and severe myocardial fibrosis. Colchicine had a protective effect on myocardium, indicated by decreased interstitial myocardial fibrosis and attenuated myocardial inflammation. It is an inflammatory cause of cardiomyopathy and myocardial fibrosis is the hallmark of this disease. Colchicine is a drug used in inflammatory diseases, and could also act on myocardial remodeling interfering in the synthesis of collagen

ELIGIBILITY:
Inclusion Criteria:

* Clinical and serological diagnosis of Chagas´disease ( Stage B1)
* Must be able to swallow tablets

Exclusion Criteria:

* myocardial infarction or coronary artery disease,
* diabetes mellitus,
* valvular disease,
* creatinine clearance <30 ml / kg / min
* contraindication to perform cardiac magnetic resonance imaging
* use of angiotensin converting enzyme inhibitors, angiotensin II receptor blockers and aldosterone blockers
* previous use of benzonidazole

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-01-05 (Estimated)

PRIMARY OUTCOMES:
Effect of colchicine on myocardial inflammation assessed by magnetic resonance imaging | 1 year
  myocardial edema quantified in grams or percent of LV mass, myocardial hyperaemia quantified in grams or percent of LV mass
Effect of colchicine on myocardial fibrosis assessed by magnetic resonance imaging | 1 year
  myocardial fibrosis quantified in grams or percent of LV mass

SECONDARY OUTCOMES:
Effect of colchicine on inflammatory markers such as interleukin-1, interleukin-6, interleukin-8, interleukin-10 | 1 year
  interleukin-1, interleukin-6, interleukin-8, interleukin-10, ELISA (pg/mL)
Effect of colchicine on inflammatory marker such as TNF-α | 1 year
  TNF-α ELISA (pg/mL)
Effect of colchicine on inflammatory marker such as interferon-gama | 1 year
  Interferon -gama ELISA (pg/mL)
Effect of colchicine on T Cruzi polymerase chain reaction | 1 year
  7500 PCR-Real time System (Life Technologies)

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Fernandes, Md, PHD, Principal Investigator — Heart Institute, University of São Paulo
Locations (1):
- Fabio Fernandes, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided